CLINICAL TRIAL: NCT06211829
Title: An Evaluation of a Antimicrobial Stewardship Recommendation Bundle for Staphylococcus Aureus Bloodstream Infections
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 016.PHA.2022.D
Record Dates: First submitted 2023-07-06; First posted 2024-01-18 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In July 2020, a bundle (Appendix C) was implemented at Methodist Dallas Medical Center where all patients with SAB were reviewed by the antimicrobial stewardship pharmacist (Monday - Friday from 0700 to 1500), a note outlining optimal interventions was written in the electronic medical record (EMR), and the recommendations were communicated to the primary team via secure messaging or telephone

DETAILED DESCRIPTION:
Evaluation of the Staphylococcus aureus bloodstream infection(SAB)bundle recommendations will allow for determination of whether this intervention is impactful and warrants the resources currently devoted to it.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age SAB during hospital admission

Exclusion Criteria:

* Patients with a history of a prior SAB during the study period (only first occurrence included)
* Blood culture collected within 48hours of patient expiring or transitioning to hospice
* Patients discharged or left before culture results were available
* Patients transferred from an outside hospital

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 18 years of age SAB during hospital admission a history of a prior SAB during the study period (only first occurrence
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
number of Staphylococcus Aureus blood stream infections (SAB) | 12 weeks
  Number of SAB occurring

SECONDARY OUTCOMES:
Number of In-hospital mortality | 12 weeks
  Number of In-hospital mortality
number of times of bacteremia | 12 weeks
  time of bacteremia
number of days of stay | 12 weeks
  duration of hospital stay
number of times of readmission | 12 weeks
  Number time of readmission
number of infection | 12 weeks
  Number of times the infection is occurring

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Holland TL, Raad I, Boucher HW, Anderson DJ, Cosgrove SE, Aycock PS, Baddley JW, Chaftari AM, Chow SC, Chu VH, Carugati M, Cook P, Corey GR, Crowley AL, Daly J, Gu J, Hachem R, Horton J, Jenkins TC, Levine D, Miro JM, Pericas JM, Riska P, Rubin Z, Rupp ME, Schrank J Jr, Sims M, Wray D, Zervos M, Fowler VG Jr; Staphylococcal Bacteremia Investigators. Effect of Algorithm-Based Therapy vs Usual Care on Clinical Success and Serious Adverse Events in Patients with Staphylococcal Bacteremia: A Randomized Clinical Trial. JAMA. 2018 Sep 25;320(12):1249-1258. doi: 10.1001/jama.2018.13155. PMID 30264119
- [Background] Perez-Rodriguez MT, Sousa A, Lopez-Cortes LE, Martinez-Lamas L, Val N, Baroja A, Nodar A, Vasallo F, Alvarez-Fernandez M, Crespo M, Rodriguez-Bano J. Moving beyond unsolicited consultation: additional impact of a structured intervention on mortality in Staphylococcus aureus bacteraemia. J Antimicrob Chemother. 2019 Apr 1;74(4):1101-1107. doi: 10.1093/jac/dky556. PMID 30689894
- [Background] Smith JR, Frens JJ, Snider CB, Claeys KC. Impact of a pharmacist-driven care package on Staphylococcus aureus bacteremia management in a large community healthcare network: A propensity score-matched, quasi-experimental study. Diagn Microbiol Infect Dis. 2018 Jan;90(1):50-54. doi: 10.1016/j.diagmicrobio.2017.10.001. Epub 2017 Oct 7. PMID 29153470
- [Background] Goto M, Schweizer ML, Vaughan-Sarrazin MS, Perencevich EN, Livorsi DJ, Diekema DJ, Richardson KK, Beck BF, Alexander B, Ohl ME. Association of Evidence-Based Care Processes With Mortality in Staphylococcus aureus Bacteremia at Veterans Health Administration Hospitals, 2003-2014. JAMA Intern Med. 2017 Oct 1;177(10):1489-1497. doi: 10.1001/jamainternmed.2017.3958. PMID 28873140
- [Background] Wenzler E, Wang F, Goff DA, Prier B, Mellett J, Mangino JE, Bauer KA. An Automated, Pharmacist-Driven Initiative Improves Quality of Care for Staphylococcus aureus Bacteremia. Clin Infect Dis. 2017 Jul 15;65(2):194-200. doi: 10.1093/cid/cix315. PMID 28379326